CLINICAL TRIAL: NCT04938362
Title: Cognitive Function and Fatigue After Brain Abscess
Status: Recruiting | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); Sunnaas Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Bjørnar Hassel, Professor, University of Oslo
Other Study IDs: Cognition/fatigue/brainabscess
Record Dates: First submitted 2021-06-13; First posted 2021-06-24 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Brain Abscess; Fatigue; Cognitive Dysfunction
MeSH Terms: conditions — Brain Abscess; Fatigue; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brain abscess patients with cognitive dysfunction and/or fatigue: This group of patients experience cognitive dysfunction and/or fatigue after brain abscess.
  Interventions: Other: FDG-PET; Other: EEG
- Brain abscess patients without cognitive dysfunction and/or fatigue: This group of patients does not experience cognitive dysfunction and/or fatigue after brain abscess.
  Interventions: Other: FDG-PET; Other: EEG

INTERVENTIONS:
Other: FDG-PET — [18F]Deoxyglucose-positron emission tomography at 0-10 years after brain abscess
Other: EEG — Electroencephalography (EEG) at 0-10 years after brain abscess

SUMMARY:
Brain abscess is a focal bacterial or fungal infection of the brain. Treatment is neurosurgical drainage of pus followed by long-term antibiotic treatment. In spite of successful treatment of the infection, long-term cognitive problems or mental fatigue may ensue. The reason for this dysfunction may be a continuing inflammatory state or damage to brain tissue caused by the abscess. The investigators will evaluate these possibilities with the use of [18F]deoxyglucose-positron emission tomography (FDG-PET) and electroencephalography (EEG) in patients who have been treated for brain abscess and who experience cognitive problems and/or fatigue. FDG-PET may identify both inflammation and altered neuronal activity (the latter indicating damage to brain tissue), and EEG may identify altered neuronal activity, including changes in neuronal network activity.

DETAILED DESCRIPTION:
Brain abscess is a focal bacterial or fungal infection of the brain, which results in a pus-filled cavity within the brain parenchyma. The incidence is approximately 1/100 000 per year, and all age groups are affected. Treatment is neurosurgical drainage of pus followed by long-term antibiotic treatment. Previously, the capsule that surrounds the pus was removed surgically; this is not usually done anymore. In spite of successful treatment of the infection, patients may experience long-lasting cognitive problems or mental fatigue. The reason for this brain dysfunction is not known.

The investigators formulated two hypotheses to explain why some patients experience long-lasting cognitive problems and/or fatigue: 1) The brain abscess caused damage to brain tissue, interrupting neuronal networks underlying cognition or 2) The abscess or the remaining capsule causes a long-lasting inflammatory state of the brain, affecting neurotransmission and cerebral function.

In this prospective study, the investigators evaluate brain abscess patients by cognitive examination by a neuropsychologist at 2 and 12 months after treatment. Participants then undergo [18F]deoxyglucose-positron emission tomography (FDG-PET). An inflammatory state in the abscess area would be identified by the FDG-PET signal. Likewise, a change in neuronal (neocortical) function would be detectable from a change in the FDG-PET signal. Participants also undergo EEG investigation to establish whether fatigue is related to alterations in EEG parameters: alpha, theta, and delta activity.

Importantly, brain damage caused by the abscess may be irreversible and functional improvement of the patient would probably have to rely on compensatory strategies, whereas an inflammatory state could probably be modified by anti-inflammatory treatment.

Further, the prognosis for the patients' cognitive problems and fatigue is probably different if the underlying cause is inflammation rather than tissue damage.

ELIGIBILITY:
Inclusion criteria:

• Patients who have completed treatment for brain abscess and who agree to participate.

Exclusion criteria:

* Patients who cannot undergo neuropsychological investigation due to unconsciousness
* Patients who cannot undergo neuropsychological investigation, being mentally too ill
* Patients who suffer from dementia
* Patients who cannot undergo FDG-PET due to claustrophobia
* Patients who cannot undergo EEG due to panic attacks
* Age under 16.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients older than 16 years, who have completed treatment for brain abscess and who agree to participate.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
A change in FDG-PET signal indicating inflammation | When all patients have been followed up for at least 1 year.
  The FDG-PET signal indicates inflammation of brain tissue or the brain abscess capsule.
A change in FDG-PET signal indicating a change in neuronal activity | When all patients have been followed up for at least 1 year.
  A change neocortical FDG-PET signal indicates a change in neuronal activity caused by brain tissue damage by the brain abscess.
A change in EEG activity indicating a change in neuronal activity based on EEG power in alpha, theta, and delta frequencies. | When all patients have been followed up for at least 1 year.
  A change neocortical EEG activity indicates a change in neuronal activity caused by brain tissue damage by the brain abscess evident as changes in EEG power in alpha, theta, and delta frequencies..

SECONDARY OUTCOMES:
Fatigue after brain abscess | When all patients have been followed up for at least 1 year.
  Neuropsychological investigation with the use of Chalder's fatigue questionnaire. Degree of fatigue is determined from the answers to 11 questions. The answer "Better than before" gives a score of 0, "Same as before" gives a score of 1, "Worse than before" gives a score of 2, and "Much worse than before" gives a score of 3. Thus, a maximum fatigue score is 33, meaning a very high degree of fatigue.
No fatigue after brain abscess | When all patients have been followed up for at least 1 year.
  Neuropsychological investigation with the use of Chalder's fatigue questionnaire. Degree of fatigue is determined from the answers to 11 questions. The answer "Better than before" gives a score of 0, "Same as before" gives a score of 1, "Worse than before" gives a score of 2, and "Much worse than before" gives a score of 3. Thus, a maximum fatigue score is 33, meaning a very high degree of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørnar Hassel, MD, PhD, Principal Investigator — University of Oslo; Daniel Dahlberg, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Patient data will be published on a group basis without identifiable characteristics. Publication will be in an international, peer-reviewed medical journal.

REFERENCES:
- [Background] Rogne AG, Muller EG, Udnaes E, Sigurdardottir S, Raudeberg R, Connelly JP, Revheim ME, Hassel B, Dahlberg D. beta-Amyloid may accumulate in the human brain after focal bacterial infection: An 18 F-flutemetamol positron emission tomography study. Eur J Neurol. 2021 Mar;28(3):877-883. doi: 10.1111/ene.14622. Epub 2020 Nov 27. PMID 33131195
- [Background] Dahlberg D, Holm S, Sagen EML, Michelsen AE, Stensland M, de Souza GA, Muller EG, Connelly JP, Revheim ME, Halvorsen B, Hassel B. Bacterial Brain Abscesses Expand Despite Effective Antibiotic Treatment: A Process Powered by Osmosis Due to Neutrophil Cell Death. Neurosurgery. 2023 Dec 12;94(5):1079-87. doi: 10.1227/neu.0000000000002792. Online ahead of print. PMID 38084989
- [Background] Hassel B, Niehusmann P, Halvorsen B, Dahlberg D. Pro-inflammatory cytokines in cystic glioblastoma: A quantitative study with a comparison with bacterial brain abscesses. With an MRI investigation of displacement and destruction of the brain tissue surrounding a glioblastoma. Front Oncol. 2022 Jul 29;12:846674. doi: 10.3389/fonc.2022.846674. eCollection 2022. PMID 35965529
- [Derived] Muller EG, Dahlberg D, Hassel B, Revheim ME, Connelly JP. Brain Abscess Causes Brain Damage With Long-Lasting Focal Cerebral Hypoactivity that Correlates With Abscess Size: A Cross-Sectional 18 F-Fluoro-Deoxyglucose Positron Emission Tomography Study. Neurosurgery. 2024 Nov 11;97(1):138-147. doi: 10.1227/neu.0000000000003268. PMID 39526777